CLINICAL TRIAL: NCT04778891
Title: The Impact of Comprehensive Medication Management Services on Clinical Outcomes in Patients With Cardiovascular Diseases at Primary Care Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zagreb (Other)
Collaborators: Health Centre Zagreb - Centre (Dom zdravlja Zagreb - Centar) (Unknown)
Responsible Party: Principal Investigator, Iva Mucalo, Associate Professor, University of Zagreb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 380-130/134-20-2
Record Dates: First submitted 2021-02-11; First posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: Cardiovascular Diseases in Old Age
Keywords: medication managements services, pharmaceutical care, primary care, elderly, control group, cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): In addition to usual care provided by general practitioner (GP) and other health care providers, a pharmacist-practitioner in collaboration with GPs from the study setting provided CMM services to patients in the intervention group. Based on the pre-defined inclusion criteria, GPs were selecting patients and referring them to the pharmacist. The individual consultation with the patient was held at the private counselling area where pharmacist and patient were able to talk face-to-face apart from the other patients. The initial assessment lasted 60-90 minutes and the follow-up evaluations 30-60 minutes. Alternatively, patients were followed-up by telephone. Communication with GPs took place in a written (electronic consultation system Health net. PRO; e-mail) and, if needed by face-to-face conversation. Each patient in the intervention group needed to agree to participate in the study by signing an Informed consent form.
  Interventions: Other: Comprehensive Medication Management services
- Control group (No Intervention): Patients in the control group received the usual care which includes GP and other health care provider visits. Data for the patients pertaining to the control group were provided by the 'control' GP and collected parallel with the intervention group. 'Control' GP profile corresponded to the profile of GPs included in the intervention group - the number of years of professional experience in the primary health care less than ten.

INTERVENTIONS:
Other: Comprehensive Medication Management services — Comprehensive Medication Management services (CMM services) is an evidence-based and patient-centred service which involves an assessment of patient's medications to determine that each medication is appropriate, effective for the medical condition being treated, safe for the patient in the presence of other medications and co-morbidities, and that the patient is able and willing to take the medications as intended. As all patient care providers need a structured, rational thought process for sound clinical decision retrieval, the Pharmacotherapy Workup was developed and adopted as a systematic problem-solving process. This process represents the cognitive work taking place in the mind of the practitioner, and is used to identify, resolve, and prevent drug therapy problems (DTP), establish therapy goals, select interventions and evaluate outcomes.
  Arms: Intervention group

SUMMARY:
Patients with established cardiovascular disease (CVD) often have multiple medications that increase the risk of prevalence of drug therapy problems (DTP), subsequently leading to unfavourable clinical and health outcomes. By providing Comprehensive Medication Management (CMM) services to patients within a healthcare system, pharmacists assess patients' medication-related needs, identify and prevent DTP, develop individualized care plan for each individual patient and evaluate and monitor outcomes. Thus, the CMM services delivered at the primary care level in collaboration with general practitioners and other healthcare providers could address this problem and by optimizing therapy improve patients' clinical outcomes and quality of life. Studies have shown that patients with chronic diseases have the greatest benefit from the CMM services. The aim of this study is to evaluate the impact of CMM services on clinical and humanistic outcomes in patients with established CVD. The study will employ prospective, longitudinal, pre- and postintervention study with a 1-year patient follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension
* Established cardiovascular disease

Exclusion Criteria:

* Organic, including symptomatic, mental disorders
* Mental and behavioural disorders due to psychoactive substance use
* Schizophrenia, schizotypal and delusional disorders
* Behavioural syndromes associated with physiological disturbances and physical factors
* Disorders of adult personality and behaviour
* Mental retardation
* Disorders of psychological development

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2021-01-17 (Actual); Study Completion 2021-01-17 (Actual)

PRIMARY OUTCOMES:
The impact of CMM services on blood pressure in elderly patients with established CVD | 1 year
  Within- and between-treatment differences for the intervention and the control group in blood pressure.

SECONDARY OUTCOMES:
The impact of CMM services on LDL cholesterol, triglycerides, HDL cholesterol and total cholesterol in elderly patients with established CVD | 1 year
  Within- and between-treatment differences for the intervention and the control group in LDL cholesterol (mmol/L), triglycerides (mmol/L), HDL cholesterol (mmol/L) and total cholesterol (mmol/L).
The impact of CMM services on health care utilization in elderly patients with established CVD | 1 year
  Between-treatment difference in the number of hospital admissions, emergency department visits and unplanned GPs visits.
The impact of CMM services on drug therapy problems in elderly patients with established CVD | 1 year
  Number and type of drug therapy problems in the intervention group.
The impact of CMM services on health related quality of life in elderly patients with established CVD assessed by EQ-5D-5L instrument. | 1 year
  Change from baseline in health related quality of life assessed by EQ-5D-5L instrument in the intervention group.
The impact of CMM services on glycated haemoglobin in elderly patients with established CVD | 1 year
  Within- and between-treatment differences for the intervention and the control group in glycated haemoglobin.

CONTACTS AND LOCATIONS:
Locations (2):
- Croatia (2):
  - Health Care Centre Zagreb - Centre, Zagreb
  - University of Zagreb Faculty of Pharmacy and Biochemistry, Zagreb

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramalho de Oliveira D, Brummel AR, Miller DB. Medication therapy management: 10 years of experience in a large integrated health care system. J Manag Care Pharm. 2010 Apr;16(3):185-95. doi: 10.18553/jmcp.2010.16.3.185. PMID 20331323
- [Background] Strand LM, Cipolle RJ, Morley PC, Frakes MJ. The impact of pharmaceutical care practice on the practitioner and the patient in the ambulatory practice setting: twenty-five years of experience. Curr Pharm Des. 2004;10(31):3987-4001. doi: 10.2174/1381612043382576. PMID 15579084
- [Background] Brummel A, Carlson AM. Comprehensive Medication Management and Medication Adherence for Chronic Conditions. J Manag Care Spec Pharm. 2016 Jan;22(1):56-62. doi: 10.18553/jmcp.2016.22.1.56. PMID 27015052
- [Background] Cranor CW, Bunting BA, Christensen DB. The Asheville Project: long-term clinical and economic outcomes of a community pharmacy diabetes care program. J Am Pharm Assoc (Wash). 2003 Mar-Apr;43(2):173-84. doi: 10.1331/108658003321480713. PMID 12688435
- [Background] Bunting BA, Smith BH, Sutherland SE. The Asheville Project: clinical and economic outcomes of a community-based long-term medication therapy management program for hypertension and dyslipidemia. J Am Pharm Assoc (2003). 2008 Jan-Feb;48(1):23-31. doi: 10.1331/JAPhA.2008.07140. PMID 18192127
- [Result] Brajkovic A, Mucalo I, Vidovic T, Gonzaga MM, Nascimento D, Balenovic A, Protrka I, De Oliveira DR. Implementation of medication management services at the primary healthcare level - a pilot study. Acta Pharm. 2019 Dec 1;69(4):585-606. doi: 10.2478/acph-2019-0055. PMID 31639091